CLINICAL TRIAL: NCT03879798
Title: A Phase I/II Study of DS-3201b, an EZH1/2 Inhibitor, in Combination With Irinotecan in Patients With Recurrent Small Cell Lung Cancer
Brief Title: DS-3201b and Irinotecan for Patients With Recurrent Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to DLTs
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-553
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Small Cell Lung Cancer
Keywords: DS-3201b; Irinotecan; 18-553
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: This study is a non-randomized phase I/II trial assessing the safety and tolerability of DS-3201b in combination with irinotecan in patients with recurrent small cell lung cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS-3201b and Irinotecan (Experimental): The first part of this study is a phase I trial to assess the safety and tolerability of DS-3201b in combination with fixed-dose irinotecan. The second part of this study will be an open label, single-arm phase II study of DS-3201b at the established recommended phase II dose (RP2D) in combination with fixed-dose irinotecan.
  Interventions: Drug: DS-3201b; Drug: irinotecan

INTERVENTIONS:
Drug: DS-3201b — 100 mg daily
Drug: irinotecan — Irinotecan 125 mg/m^2 intravenously on days 1 and 8 every 3 weeks in a 21-day cycle.

SUMMARY:
This study will test the safety of the study drug, DS-3201b, given in combination with irinotecan to people who have recurrent small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Ability to comply with the study protocol as per the investigator's judgment
* Age ≥ 18 years at the time of signing the ICF
* Life expectancy ≥ 12 weeks
* Karnofsky performance status ≥ 70% or ECOG 0, -1 or 2
* Pathologically confirmed diagnosis of small cell lung cancer. Patients with a diagnosis of combined small cell lung cancer with other histologies may be considered for inclusion if the predominant histology is SCLC and only after discussion with the study PI. Patients with transformed SCLC from NSCLC are allowed on study after discussing with the MSKCC or JHU Study PI
* Radiographically documented progression of disease after prior treatment with a platinum doublet regimen. Patients who received a platinum doublet regimen in combination with immunotherapy are still eligible for the study.
* Measurable disease according to RECIST v1.1
* Adequate tissue sample available for both IHC testing of IHC testing of SLFN11 and H3K27me3 and molecular profiling (archived tissue block or 20 unstained slides). Tissue sample can be either from an initial pre-platinum-based chemotherapy sample OR from a repeat biopsy sample after progression on platinum-based chemotherapy.
* Concurrent consent to the appropriate biospecimen research protocols at MSKCC (#06-107 Storage and Research Use of Human Biospecimens) and at JHU.
* Adequate hematologic and end-organ function, as defined by the following laboratory test results obtained within 14 days prior to initiation of study treatment:

  °Adequate bone marrow function as defined by:
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1500/µL) without granulocyte colony-stimulating factor support within 2 weeks prior to starting study therapy
  * Hemoglobin ≥ 9 g/dL (transfusions to meet this criterion are allowed)
  * Platelets ≥ 150 x 10^9/L without transfusion
* Adequate renal function as defined by:

  °Creatinine clearance ≥ 50 mL/min as calculated using the modified Cockcroft-Gault equation or Modification of Diet in Renal Disease (MDRD) formula OR serum creatinine ≤1.5 x ULN
* Adequate hepatic function as defined by:

  * AST, ALT, and alkaline phosphatase (ALP) ≤ 3 x ULN with the following exceptions
  * Patients with documented liver metastases: AST, ALT and ALP ≤ 5 x ULN
  * Total bilirubin ≤ 2.0 mg/dL
  * For patients not receiving therapeutic anticoagulation:
  * stable anticoagulant regimen
  * INR ≤ 1.5 x ULN
  * aPTT ≤ 1.5 x ULN
* Patients with baseline clinical symptoms or laboratory abnormalities that do not meet the definition of dose-limiting toxicity (DLT).
* Nonsterilized female patients of reproductive age group and male patients should use highly effective methods of contraception through defined periods during and after study treatment as specified below:

  * Female patients must meet 1 of the following:
  * Postmenopausal for at least 1 year before the screening visit, or
  * Surgically sterile, or
  * If she is of childbearing potential, agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * Female patients must agree to not donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Examples of highly effective contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, and established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to

    1. of the following:
  * Practice highly effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or
  * Practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * Male patients must agree to not donate sperm during the course of this study or 6 months after receiving their last dose of study drug(s).
  * Patient is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.

Exclusion Criteria:

* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.
* Untreated CNS metastases
* Patients with treated CNS metastases are allowed on the study as long as their clinical symptoms are adequately controlled and the daily dose of steroid use is equivalent to or less than 10 mg of prednisone.
* Is receiving concomitant treatment with a strong inhibitor or inducer of CYP3A4/5 within 7 days of first receipt of DS-3201b.

  °Consumption of herbs/fruits that may have an influence on PK of DS-3201b (strong CYP3A inhibitors or inducers) such as St. John's wort, star fruit, Seville orange or Seville orange-containing foods and beverages, grapefruit or grapefruit-containing food or beverages should be avoided from 14 days prior to the start of the study and throughout the entire study.
* Prior exposure to DS-3201b or other inhibitors of enhancer of zeste homologue-2 (EZH2)
* Prior exposure to topoisomerase inhibitors, including topotecan and irinotecan

  * Refractory nausea and vomiting, malabsorption, biliary shunt, significant bowel resection, or any other condition that significantly affects gut motility or absorption and would preclude adequate absorption of DS-3201b in the opinion of the treating physician and/or PI.
  * Currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks prior to the initiation of study treatment. Anticancer therapies include chemotherapy, biologics, targeted therapies, immunologics, or other investigational therapy.
* Currently receiving radiation therapy, or who have received radiation within 2 weeks prior to the initiation of study treatment.
* Patients who have not recovered to Grade ≤1 or baseline from adverse events due to prior anticancer therapy.
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).

  * NOTE: Procedures such as a percutaneous biopsy, pleural catheter insertion, placement of a central venous catheter or other minor procedures are permitted.
  * Uncontrolled or significant cardiovascular disease, including the following:
  * Evidence of prolongation of QT/QTc interval (e.g., repeated episodes of QT corrected for heart rate using Fridericia's method [QTcF] >450 ms for men and >470 ms for females) ECG from 12-lead electrocardiogram for measurement of corrected QT interval according to the Fridericia formula: electrocardiogram must be registered at rest. For any EKG assessment, if the initial EKG shows a prolonged QTc, then two additional EKGs will be obtained, resulting in three specimens taken after a space of

    1 minute, and the mean of the 3 EKGs will be used to determine eligibility and for grading of TRAEs.
  * Diagnosed or suspected long QT syndrome, or known family history of long QT syndrome
  * History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes
  * Uncontrolled arrhythmia (subjects with asymptomatic, controllable atrial fibrillation may be enrolled), or asymptomatic persistent ventricular tachycardia
  * Subject has clinically relevant bradycardia of <50 bpm unless the subject has a pacemaker
  * History of second- or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers, and have no history of fainting or clinically relevant arrhythmia with pacemakers, within 6 months prior to Screening
  * Myocardial infarction within 6 months prior to Screening
  * Angioplasty or stent graft implantation within 6 months prior to Screening
  * Uncontrolled angina pectoris within 6 months prior to Screening
  * New York Heart Association (NYHA) Class 3 or 4 congestive heart failure
  * Coronary/peripheral artery bypass graft within 6 months prior to Screening
  * Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) Complete left or right bundle branch block
* Patients who are currently taking medications that are known to prolong the QT interval and are clearly associated with a known risk of Torsades de Pointes (TdP) even when taken as recommended. Please see Section 11.6 for a full list of excluded medications. Patients who are able to discontinue any prohibited medication prior to the start of study drug at Day -7 will still be considered eligible for the study.
* Have a known hypersensitivity to any of the components of or known hypersensitivity to either the study drug itself or any of the inactive ingredients in the study drug product.
* Known liver cirrhosis.
* Uncontrolled active infection requiring IV antibiotic, antiviral, or anti-fungal medications within 14 days prior to initiation of study treatment.

  °Infections controlled on concurrent anti-microbial agents and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Congenital or acquired immunodeficiency, including patients with known history or infection with human immunodeficiency virus (HIV).

  °NOTE: HIV-positive patients who are taking anti-retroviral therapy are still ineligible due to potential PK interactions with DS-3201b.
* Active tuberculosis
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test Hepatitis B testing (HBV surface antigen and core antibody) is required only if not done previously

  °Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test, are eligible for the study. Hepatitis B testing is required only if not done previously
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test. Hepatitis C testing (HCV antibody) is required only if not done previously

  °The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Female patients who have a positive serum pregnancy test during screening or a positive urine pregnancy test on Day 1 before first dose of study drug.
* Female patients who are lactating and/or plan to breastfeed during the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose Level 1: Dose Level 1 (DS-3201b 100mg)
- Phase I, Dose Level 2: Dose Level 2 (DS-3201b 150mg)
- Phase I, Dose Level 3: Dose Level 3 (DS-3201b 200mg)
- Phase I, Dose Level 4: Dose Level 4 (DS-3201b 250mg)
- Phase I, Dose Level 5: Dose Level 5 (DS-3201b 300mg)
- Phase 2: DS-3201b 100mg
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase I, Dose Level 5 | Phase 2
Started | 6 | 6 | 0 | 0 | 0 | 10
Completed | 6 | 6 | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were not treated at Dose Level 3, 4 or 5
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase I, Dose Level 5 | Phase 2 | Total
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 10 | 22
Age, Continuous [Median (Full Range); unit: years] | 72 [60 to 79] | 59 [44 to 70] |  |  |  | 67 [44 to 79] | 66 [44 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 |  |  |  | 7 | 13
  Male | 3 | 3 |  |  |  | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 |  |  |  | 0 | 1
  Not Hispanic or Latino | 5 | 5 |  |  |  | 0 | 10
  Unknown or Not Reported | 1 | 0 |  |  |  | 10 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  |  | 0 | 0
  Asian | 0 | 0 |  |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0 | 0
  Black or African American | 0 | 0 |  |  |  | 2 | 2
  White | 6 | 6 |  |  |  | 7 | 19
  More than one race | 0 | 0 |  |  |  | 0 | 0
  Unknown or Not Reported | 0 | 0 |  |  |  | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 |  |  |  | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase l) of DS-3201/Valemetostat
Description: Will employ a standard 3-by-3 dose-escalation phase I study design to investigate the maximum tolerated dose (MTD) of DS-3201b/valemetostat in combination with fixed dose irinotecan. The study population for Phase I dose-escalation will include only patients who complete at least 1 full cycle of treatment (including the initial 7-day safety run-in and the complete 21-days of Cycle 1); only these patients will be considered evaluable for DLT and determination of the MTD.
Time Frame: 1 year
Population: MTD determined from phase I
Measure: Number; unit: mg
Groups:
- All Phase I Participants, Dose Level 1 & Dose Level 2: Dose Level 1 (DS-3201b 100mg)
  Dose Level 2 (DS-3201b 150mg)
- Phase 2: The first part of this study is a phase I trial to assess the safety and tolerability of DS-3201b in combination with fixed-dose irinotecan. The second part of this study will be an open label, single-arm phase II study of DS-3201b at the established recommended phase II dose (RP2D) in combination with fixed-dose irinotecan. Dose-Escalation, which enrolled a total of 12 patients at MSK, is completed. Phase 1 of this study determined that the highest and safest dose of DS-3201b in patients was 100 mg daily.
  DS-3201b: 100 mg daily
  irinotecan: Irinotecan 125 mg/m^2 intravenously on days 1 and 8 every 3 weeks in a 21-day cycle.
Arm/Group | All Phase I Participants, Dose Level 1 & Dose Level 2 | Phase 2
Number analyzed (Participants) | 10 | 0
mg | 100 |

2. Primary Outcome: Objective Response Rate (ORR) (Phase II)
Description: The Response Evaluation Criteria in Solid Tumors Group (RECIST v1.1) criteria will be used to evaluate the response to treatment
Time Frame: 1 year
Population: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Measure: Number (95% Confidence Interval); unit: % of participants
Groups:
- Phase I: The first part of this study is a phase I trial to assess the safety and tolerability of DS-3201b in combination with fixed-dose irinotecan.
- Phase 2: The second part of this study will be an open label, single-arm phase II study of DS-3201b at the established recommended phase II dose (RP2D) in combination with fixed-dose irinotecan.
Arm/Group | Phase I | Phase 2
Number analyzed (Participants) | 0 | 10
% of participants |  | 21 [6 to 46]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants were not treated on Dose Level 3, 4 or 5
Groups:
- Phase I, Dose Level 1: Dose Level 1: 100mg
- Phase I, Dose Level 2: Dose Level 2: 150mg
- Phase I, Dose Level 3: Dose Level 3: 200mg
- Phase I, Dose Level 4: Dose Level 4: 250mg
- Phase I, Dose Level 5: Dose Level 5: 300mg
- Phase 2: Dose Level 2: 100mg
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase I, Dose Level 5 | Phase 2
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/6 | 0/0 | 0/0 | 0/0 | 8/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/0 | 0/0 | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 0/0 | 0/0 | 0/0 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose Level 1 (N=6) | Phase I, Dose Level 2 (N=6) | Phase I, Dose Level 3 (N=0) | Phase I, Dose Level 4 (N=0) | Phase I, Dose Level 5 (N=0) | Phase 2 (N=10)
Diarrhea (Gastrointestinal disorders) | 5 | 4 | NA | NA | NA | 6
Fatigue (General disorders) | 3 | 4 | NA | NA | NA | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | NA | NA | NA | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | NA | NA | NA | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | NA | NA | NA | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | NA | NA | NA | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | NA | NA | NA | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | NA | NA | NA | 1
Dizziness (Nervous system disorders) | 1 | 1 | NA | NA | NA | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | NA | NA | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03879798/Prot_SAP_000.pdf